CLINICAL TRIAL: NCT04286919
Title: The Heat Is On To Increase Physical Activity: Comparing Two Different Methods To Prescribe Exercise
Brief Title: Comparing Two Different Methods to Prescribe Exercise
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Linda Pescatello, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H18-266
Record Dates: First submitted 2020-02-20; First posted 2020-02-27 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Physical Activity; Health Behavior
Keywords: Exercise; Adherence
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with 1 control group and 1 intervention group. The control group is getting the standard of care exercise prescription based on the 2018 physical activity guidelines for Americans and the intervention group is getting a new method of prescribing exercise based on new research informing the 2018 Move Your Way initiative where all physical activity across all types and intensities is advised.
Who Masked: Participant
Masking Description: Participants do not know that there is another group getting a different exercise prescription. At the end of their participation, all participants will be offered the other exercise prescription.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ExRx#1: Physical Activity Guidelines (Active Comparator): ExRx#1 uses the Frequency, Intensity, Time, and Type or FITT principle of exercise prescription to prescribe the Physical Activity Guidelines for Americans which is a weekly goal of 150-minutes of moderate intensity aerobic physical activity plus 2 days of muscle strengthening physical activity. ExRx#1 communicates the ultimate goal of the physical activity guidelines for Americans using an image adopted from the physical activity guidelines website that depicts the weekly goal. There are 12 weeks of exercise guidelines that will progress participants from being physically inactive to meeting the physical activity guidelines ultimate weekly goal by providing a weekly prescription of Frequency, Intensity, Time, and Type of physical activity that accomplishes meeting the physical activity guidelines weekly goal.
  Interventions: Behavioral: A Randomized Controlled Trial Comparing the Physical Activity Guidelines for Americans to a New Method of Exercise Prescription Among College Students
- ExRx#2: Heat Map (Experimental): ExRx#2 uses the heat map image published in the 2018 Physical Activity Guidelines Advisory Committee Scientific Report that communicates the dose-response relationship between increased physical activity and improved health to prescribe the message that all physical activity across all Frequencies, Intensities, Time bouts and Types (FITT) counts towards health. ExRx#2 is founded in the Integrated Behavior Change Theory and emphasizes that all physical activity matters regardless of FITT as depicted by the heat map image. There are 12 weeks of exercise guidelines that will progress participants from being physically inactive to meeting the ExRx#2 heat map ultimate weekly goal of moving more throughout the day across all intensities in order to achieve optimal health as represented by the deep green color on the bottom right of the heat map image.
  Interventions: Behavioral: A Randomized Controlled Trial Comparing the Physical Activity Guidelines for Americans to a New Method of Exercise Prescription Among College Students

INTERVENTIONS:
Behavioral: A Randomized Controlled Trial Comparing the Physical Activity Guidelines for Americans to a New Method of Exercise Prescription Among College Students — A randomized controlled trial comparing the 2018 Physical Activity Guidelines for Americans weekly recommendations of 150-minutes of moderate intensity physical activity plus 2 days of muscle-strengthening physical activity to the Move Your Way Campaign message of increasing any and all physical activity to accumulate more movement throughout the week across all types and intensities.
  Other Names: Comparing the Physical Activity Guidelines for Americans to The Move Your Way Campaign Methods of Exercise Prescription Among College Students

SUMMARY:
Practical interventions are needed to increase physical activity (PA) levels in insufficiently active individuals. HEAT is a randomized controlled trial comparing two different exercise prescription (ExRx) methods to increase PA volume among insufficiently active UConn students. Students will be randomized to two groups: (1) ExRx#1 will emphasize meeting the Physical Activity Guidelines for Americans via the Frequency, Intensity, Time, and Type or FITT principle of ExRx; and (2) ExRx#2 will be founded in the Integrated Behavior Change Theory and based on the 2018 Physical Activity Guidelines Review Committee Scientific Report heat map which emphasizes that all PA counts. HEAT aims to assess the effectiveness of each ExRx individually and comparatively to one another for each outcome measure. We hypothesize that UConn students in ExRx#2 will increase PA volume more than ExRx#1 in response to the 12wk ExRx due to its foundation in the IBC. If our hypothesis proves correct we aim to inform healthcare providers on university campuses on which method of ExRx is more effective at increasing PA participation among their insufficiently active students.

DETAILED DESCRIPTION:
Being regularly physically active, defined as exercising at least 3-days/wk for 30-min provides essential and seemingly unlimited health benefits. To emphasize the importance of the health benefits of physical activity (PA), the United States government recently provided us with The Physical Activity Guidelines for Americans (PAG) 2nd edition. This recommended PA prescription for improving and maintaining health includes 150-min/wk of moderate intensity aerobic PA plus 2-days of muscle-strengthening PA. Yet, an estimated 26% of American adults and 36% of college students do not perform any leisure-time PA. A novelty of the PAG 2nd edition is the updated research acknowledging that PA exists on a spectrum where any and all movement is beneficial to health. This update emphasizes that the steepest decrease in relative risk of all-cause mortality among physically inactive individuals occurs with the substitution of sedentary behavior for light intensity movement, inherently encompassing lifestyle activities as healthy, meaningful PA. The 2018 Physical Activity Guidelines Advisory Committee Scientific Report (PAGACSR) conceptualizes this important public health message with the creation of a heat map relating PA with all-cause mortality, creatively depicting the dose-response effect of increased PA on health. The Office of Disease Prevention and Health Promotion contends that this new emphasis on all PA counting towards health can serve as a method of increasing PA in physically inactive individuals as demonstrated by the launch of the Move Your Way initiative. The all movement counts message can encompass the Integrated Behavior Change Theory (IBC) which attributes increased PA to perceived behavioral control due to higher autonomy.

HEAT is a Randomized Controlled Trial (RCT) comparing the PAG exercise prescription (ExRx#1) of 150-min/wk of moderate intensity aerobic PA plus 2-days of muscle-strengthening PA to a new method of exercise prescription (ExRx) using the everything counts message depicted by the heat map (ExRx#2) to prescribe exercise to physically inactive individuals. ExRx#1 uses the Frequency, Intensity, Time, and Type or FITT principle of ExRx to relay the PAG; and ExRx#2 will be founded in the Integrated Behavior Change Theory (IBC) and emphasize that all PA counts to relay the message of the heat map. ExRx#1 communicates the PAG ultimate weekly goal ExRx using an image adopted from the PAG website that depicts the 150-minutes of aerobic and 2 days of muscle strengthening exercise and provides a weekly prescription on the FITT of how to accomplish this weekly goal. ExRx#2 uses the heat map image to communicate the ExRx of all movement counts and that exercise can be done along any FITT.

Both ExRx were created by an expert panel of exercise professionals including the principal investigator Linda S Pescatello, PhD, who was senior editor of the American College of Sports Medicine Guidelines for Exercise Testing and Prescription 9th edition and one of the 17 Advisory Committee members of the PAGACSR which provided the scientific foundation for the PAG 2nd edition.

1. ExRx #1: The ExRx given to participants each week represents the ultimate weekly goal of 150-min of aerobic PA plus 2-days of muscle-strengthening PA to support optimal health. For example, the ExRx on week 6 suggests 3-days/wk of 50-min of aerobic PA plus 2-days of 30-min of muscle-strengthening PA in the form of resistance or neuromotor exercise. The ExRx then gives examples of taking a 50-min moderate intensity Zumba class on one day to fulfill part of the weekly aerobic PA guideline and 2-3 sets of 8-12 reps of resistance exercises for 30-min of muscle-strengthening PA on another day.
2. ExRx #2: The ExRx given to participants each week represents the ultimate weekly goal of moving more throughout the day across all intensities in order to achieve optimal health as represented by the deep green color on the bottom right of the heat map image that represented high amounts of activity and good health. For example, the ExRx on week 6 suggests including a variety of moderate intensity physical activities and light intensity physical activities to achieve the deep green color on the bottom right of the heat map. The ExRx then gives the examples of taking a Zumba class and weight training.

Subjects will be randomly assigned to receiving either ExRx#1 (n=30), or ExRx#2 (n=30). All subjects will participate in a 12-week unsupervised ExRx program that will safely progress them from being physically inactive to becoming physically active. Each week subjects of both groups will be sent an ExRx in the form of PA recommendations for the week that will be matched in terms of intervention setting, behavior change strategies, mode of intervention delivery, suggestions for types of PA to do, action planning, goal timeframe, and feedback. The difference between the two ExRx methods is the messaging of the specific frequency, intensity time, and type to follow in ExRx#1 versus giving only suggestions of exercises to do and no frequency, intensity, time or type restriction as "all movement counts" is emphasized in ExRx#2. Both groups will be given the main goal of the guidelines they are randomized to along with the same information on the definitions of aerobic, resistance, neuromotor, flexibility and concurrent exercise along with how to measure intensity of PA using the talk test and the Borg Ratings of Perceived Exertion 6-20 scale. Each participant will be verbally explained the overall goal of the ExRx and walked through the definitions to ensure complete understanding of each mode of PA and how to monitor intensity of activity. Both groups will be instructed that the guidelines will progress them from being physically inactive to meeting the overall goal of the ExRx from weeks 1-6; then the guidelines will stay consistent in prescribing the overall goal of the ExRx from weeks 6-12. In both groups, the ExRx is described as effective for improving and maintaining health and that all PA participation is at their own discretion and they can do whatever PA type they would like. Participants in both groups will be given the same exercise compendium of aerobic and resistance exercises to choose from in case they are unsatisfied with the example types of PA recommended in the weekly guidelines. Researchers will stress the goal of accurately recording PA and exercise regardless of if the recommendations given to them are met or not.

Currently 36% of University students are physically inactive. Due to barriers such as lack of time, exercising 150-min/wk+ and accomplishing a specific FITT such as the ExRx#1 provides may seem unattainable. In contrast, the ExRx#2 demonstrates a simple message to move more however you can, allowing for practical uptake of increased PA and using the IBC to connect the intention to exercise with the behavior through increased self-efficacy and autonomy. We hypothesize that ExRx #2 will elicit greater increases in PA volume from baseline (BL) to post-test at the end of the 12 weeks of guidelines (12W) compared to ExRx#1. We hypothesize that ExRx#2 will produce greater improvement in autonomy and self-efficacy compared to ExRx#1 at 12W.

Anthropometrics, health-fitness assessments, PA tracking and questionnaires will be administered at BL, 6W and 12W. All questionnaires will be administered in person using Qualtrics Secure encrypted database and will be compared between groups at BL, 6W and 12W to measure changes over time. Age will be assessed in years. Height (cm) and weight (kg) will be measured and used to calculate body mass index in m2/kg. Waist circumference will be measured at the height of the iliac crest with a Gulick tape measure in cm. Cardiorespiratory fitness will be assessed using a modified and validated Harvard Step Test protocol where participants step up and down on a 30cm box at a rate of 30 steps/min for 3-min and recovery heart rate (HR) is recorded. Muscular endurance will be measured via the push-up test with males performing repetitions until failure in the standard position and females in the modified kneeling position. Handgrip strength is a validated measure of overall muscular strength and will be measured using a validated protocol in the dominant hand with the Jamar Hydraulic Handgrip Dynamometer. Flexibility will be measured in cm using a Sit and Reach Flexibility Box. Timeline Follow-Back for Exercise (TLFB-E) is a self-report calendar diary method for logging daily exercise and PA, and sitting and sleeping time. Participants will record daily PA frequency, type, duration (min) and intensity using the Borg 6-20 scale. Researchers will assess the TLFB-E weekly to ensure students are actively participating in reading the ExRx guidelines and logging activity. Paffenbarger Physical Activity Questionnaire Question 8 will measure duration (min) in each intensity of PA plus time spent sleeping and sitting for a typical weekday and weekend day. PA volume will be calculated in MET.min/wk. Actical® accelerometers will be given to participants to wear on their hip for 4 consecutive days including 2 weekdays and 2 weekend days as an objective measure of PA volume in MET.min/day, steps/day and time spent in light, moderate and vigorous intensities. Transtheoretical Model Stage of Change will assess readiness to take action to exercise regularly and measures transitions in this readiness. Motivation for Physical Activity will determine type of motivation for PA (e.g., intrinsic vs external) and self-perceived autonomy. Marcus Self-Efficacy questionnaire will measure confidence for exercising when 5 different perceived barriers present. Task Self-Efficacy will measure confidence for exercising 3 times/wk at increasing durations. Barriers to Self-Efficacy will assess confidence in exercising 3days/wk for the next 3 months in the presence of possible barriers to exercise.

Group descriptive statistics will be presented as mean±standard deviation and ANOVA will be performed to determine if there are BL differences between the groups. All BL, 6W and 12W measures of PA and the psychosocial questionnaires will be analyzed with repeated measures ANCOVA using gender as a fixed factor and age, BMI, WC and other baseline descriptive characteristics as possible covariates. Post-hoc analyses will be used to test differences in groups and for 3 time points if there are significant time, group or time*group interactions. Methods such as multiple imputation and estimated means algorithm will be used to carry out statistical inferences in the presence of missing data. All analyses will be set at the alpha level of .05 and will be carried out using SPSS Version 25.

ExRx #1 utilizes the widely-used gold standard FITT principle of ExRx to promote achieving the PAG. ExRx #2 uses updated research on the benefits of light intensity movement and the all movement counts message founded in the IBC to inherently support autonomy and higher self-efficacy to connect the intention to exercise with the behavior. This RCT will inform practitioners about which message resonates more with physically inactive students so we can more effectively promote healthy, active lifestyles.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old.
* Participants will attend UConn Storrs campus as an undergraduate or graduate student during the study.
* Participants must be physically inactive as defined by participating in less than or equal to 2 days of planned, structured physical activity over the past 12 weeks.
* Any and all races may be included.
* Participants will be healthy with no diagnosed cardiovascular, pulmonary, metabolic, or other chronic diseases or depression and not taking medication for any of these chronic diseases or health conditions as defined by answering "no" to all General Health Questions listed in the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+).
* Anyone scoring less than a 19 on the Beck Depression Inventory.
* Those who answer "yes" to 3 or less on the eating questionnaire will be included.
* Between 18-35 m2/kg.
* Participants should be non-smokers for at least 6 months prior to entry.
* Participants should drink <2 alcoholic drinks daily.
* Women who are not pregnant or lactating and do not plan on becoming pregnant.
* Participants with no arthritis or orthopedic problems inhibiting their ability to exercise across all intensities without exacerbating the problem.
* Participants willing to maintain their habitual diet throughout the study.
* Participants wanting to enter the study for reasons that do not include weight loss.
* Participants should be willing and able to consent to all data collection processes including the intended timeline of the study procedures as well as all questionnaires, fitness assessments, and physical activity monitor usage.
* Participants who are willing to use only the physical activity program given to them by researchers and are willing to refrain from obtaining and using another program given to them by anyone else besides study researchers. Participants must also agree to not look at the physical activity guidelines being administered to the other intervention group that they are not assigned to.

Exclusion Criteria:

* <18 years old
* Not attending UConn Storrs campus during the duration of their enrollment.
* Answering "no" to any question on the 12-item checklist of inclusion criteria
* Participating in more than 2 days of planned, structured physical activity over the past 12 weeks.
* Unhealthy students as determined by answering "yes" to any question listed on the PAR-Q+.
* Scoring a 19 or higher on the Beck Depression Inventory.
* Those who answer "yes" to more than 3 statements on the SCOFF eating disorder questionnaire will be excluded.
* BMI <18 or >35 m2/kg.
* People who currently smoke, plan on smoking or have smoked tobacco within the last 6 months.
* People drinking 2 or more alcoholic drinks daily.
* Women who are pregnant or lactating.
* People with arthritis or orthopedic problems will not be enrolled if these conditions compromise their completion of the exercise protocols or ability to exercise across all intensities.
* People unwilling to maintain their habitual diet as we request throughout study participation.
* We will not recruit subjects whose primary motivation for enrolling is to lose weight.
* People who do not think they will be able to complete all study protocols at the times they are scheduled to complete them. This includes the completion of study time logs and all study visits.
* Anyone not willing to confirm that they will refrain from obtaining another exercise program or viewing that of the other group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Physical Activity Volume change from Baseline to 12 weeks | 12 weeks
  Actical® (Mini Meter, Respironics Inc.) accelerometers will be given to participants to wear on their hip for 4 consecutive days including 2 weekdays and 2 weekend days as an objective measure of PA volume in MET-hours/day. This data will be collected at baseline before the exercise guidelines start and at week 12 of the exercise guidelines to measure change from baseline to 12 weeks.

SECONDARY OUTCOMES:
Autonomy Score Change from Baseline to 12 weeks | 12 weeks
  Motivation for Physical Activity will be assessed by a questionnaire developed using the Self-Determination theory which is found to be valid and reliable in assessing type of motivation for PA in adults. This instrument has 16 items that will allow researchers to determine type of motivation (e.g., intrinsic versus external) and create a relative autonomy index for each subject as a direct result of the scoring of this questionnaire. This score is used to detect level of autonomy in exercise. This measure will be administered at baseline and 12 weeks to measure change from baseline over 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Linda S Pescatello, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. All data will be analyzed and presented in aggregate as accepted by the University of Connecticut IRB.

REFERENCES:
- [Background] Powell KE, King AC, Buchner DM, Campbell WW, DiPietro L, Erickson KI, Hillman CH, Jakicic JM, Janz KF, Katzmarzyk PT, Kraus WE, Macko RF, Marquez DX, McTiernan A, Pate RR, Pescatello LS, Whitt-Glover MC. The Scientific Foundation for the Physical Activity Guidelines for Americans, 2nd Edition. J Phys Act Health. 2018 Dec 17:1-11. doi: 10.1123/jpah.2018-0618. Online ahead of print. PMID 30558473
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Riebe D, Ehrman J, Liquori G, Magal M. ACSM's Guidelines for Exercise Testing and Prescription tenth edition. 10th ed. Wolters Kluwer: Katie Feltman; 2018.
- [Background] Hagger MS, Chatzisarantis NL. An integrated behavior change model for physical activity. Exerc Sport Sci Rev. 2014 Apr;42(2):62-9. doi: 10.1249/JES.0000000000000008. PMID 24508739
- [Background] Williams SL, French DP. What are the most effective intervention techniques for changing physical activity self-efficacy and physical activity behaviour--and are they the same? Health Educ Res. 2011 Apr;26(2):308-22. doi: 10.1093/her/cyr005. Epub 2011 Feb 14. PMID 21321008
- [Background] Samdal GB, Eide GE, Barth T, Williams G, Meland E. Effective behaviour change techniques for physical activity and healthy eating in overweight and obese adults; systematic review and meta-regression analyses. Int J Behav Nutr Phys Act. 2017 Mar 28;14(1):42. doi: 10.1186/s12966-017-0494-y. PMID 28351367
- [Background] Chatzisarantis NL, Hagger MS, Smith B. Influences of perceived autonomy support on physical activity within the theory of planned behavior. European Journal of Social Psychology 2007;37(5):934-954.
- [Background] Keating XD, Guan J, Pinero JC, Bridges DM. A meta-analysis of college students' physical activity behaviors. J Am Coll Health. 2005 Sep-Oct;54(2):116-25. doi: 10.3200/JACH.54.2.116-126. PMID 16255324
- [Background] Trost SG, Owen N, Bauman AE, Sallis JF, Brown W. Correlates of adults' participation in physical activity: review and update. Med Sci Sports Exerc. 2002 Dec;34(12):1996-2001. doi: 10.1097/00005768-200212000-00020. PMID 12471307
- [Background] Hill LS, Reid F, Morgan JF, Lacey JH. SCOFF, the development of an eating disorder screening questionnaire. Int J Eat Disord. 2010 May;43(4):344-51. doi: 10.1002/eat.20679. PMID 19343793
- [Background] Simpson K, Parker B, Capizzi J, Thompson P, Clarkson P, Freedson P, Pescatello LS. Validity and reliability question 8 of the Paffenbarger Physical Activity Questionnaire among healthy adults. J Phys Act Health. 2015 Jan;12(1):116-23. doi: 10.1123/jpah.2013-0013. Epub 2014 Apr 11. PMID 24733349
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Ibrahim JG, Chen M, Lipsitz SR, Herring AH. Missing-data methods for generalized linear models: A comparative review. Journal of the American Statistical Association 2005;100(469):332-346.
- [Background] Rubin DB. Inference and missing data. Biometrika 1976;63(3):581-592.
- [Background] American Society of, Hand Therapists. Clinical assessment recommendations. 1992.
- [Background] KEEN EN, SLOAN AW. Observations on the Harvard step test. J Appl Physiol. 1958 Sep;13(2):241-3. doi: 10.1152/jappl.1958.13.2.241. No abstract available. PMID 13575336
- [Background] Panza GA, Weinstock J, Ash GI, Pescatello LS. Psychometric Evaluation of the Timeline Followback for Exercise among College Students. Psychol Sport Exerc. 2012 Nov;13(6):779-788. doi: 10.1016/j.psychsport.2012.06.002. Epub 2012 Jun 20. PMID 22844226
- [Background] Matthews CE, Ainsworth BE, Thompson RW, Bassett DR Jr. Sources of variance in daily physical activity levels as measured by an accelerometer. Med Sci Sports Exerc. 2002 Aug;34(8):1376-81. doi: 10.1097/00005768-200208000-00021. PMID 12165695
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] McAuley E, Courneya KS. The subjective exercise experiences scale (SEES): Development and preliminary validation. Journal of Sport and Exercise Psychology 1994;16(2):163-177..
- [Background] Resnick B, Zimmerman SI, Orwig D, Furstenberg AL, Magaziner J. Outcome expectations for exercise scale: utility and psychometrics. J Gerontol B Psychol Sci Soc Sci. 2000 Nov;55(6):S352-6. doi: 10.1093/geronb/55.6.s352. PMID 11078112
- [Background] Deci E. Exercise Self-Regulation Questionnaires. Self-Determination Theory: An Approach to Human Motivation and Personality- The Self-Regulation Questionnaires 2004.
- [Background] McAuley E. The role of efficacy cognitions in the prediction of exercise behavior in middle-aged adults. J Behav Med. 1992 Feb;15(1):65-88. doi: 10.1007/BF00848378. PMID 1583674
- [Background] McAuley E, Blissmer B. Self-efficacy determinants and consequences of physical activity. Exerc Sport Sci Rev. 2000 Apr;28(2):85-8. PMID 10902091
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Marcus, B H and Forsyth L H. Motivating People to Be Physically Active. : Human Kinetics; 2003. p. 21.
- [Background] O'Brien E, Beevers G, Lip GY. ABC of hypertension: Blood pressure measurement. Part IV-automated sphygmomanometry: self blood pressure measurement. BMJ. 2001 May 12;322(7295):1167-70. doi: 10.1136/bmj.322.7295.1167. No abstract available. PMID 11348915
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves JW, Hill MN, Jones DH, Kurtz T, Sheps SG, Roccella EJ; Council on High Blood Pressure Research Professional and Public Education Subcommittee, American Heart Association. Recommendations for blood pressure measurement in humans: an AHA scientific statement from the Council on High Blood Pressure Research Professional and Public Education Subcommittee. J Clin Hypertens (Greenwich). 2005 Feb;7(2):102-9. doi: 10.1111/j.1524-6175.2005.04377.x. No abstract available. PMID 15722655
- [Background] Roshanaei-Moghaddam B, Katon WJ, Russo J. The longitudinal effects of depression on physical activity. Gen Hosp Psychiatry. 2009 Jul-Aug;31(4):306-15. doi: 10.1016/j.genhosppsych.2009.04.002. Epub 2009 May 13. PMID 19555789
- [Background] Beck AT, Steer RA, Carbin MG. Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clin Psychol Rev 1988;8(1):77-100.
- [Background] Morgan JF, Reid F, Lacey JH. The SCOFF questionnaire: assessment of a new screening tool for eating disorders. BMJ. 1999 Dec 4;319(7223):1467-8. doi: 10.1136/bmj.319.7223.1467. No abstract available. PMID 10582927
- [Background] Bravata DM, Smith-Spangler C, Sundaram V, Gienger AL, Lin N, Lewis R, Stave CD, Olkin I, Sirard JR. Using pedometers to increase physical activity and improve health: a systematic review. JAMA. 2007 Nov 21;298(19):2296-304. doi: 10.1001/jama.298.19.2296. PMID 18029834
- [Background] McEwan D, Harden SM, Zumbo BD, Sylvester BD, Kaulius M, Ruissen GR, Dowd AJ, Beauchamp MR. The effectiveness of multi-component goal setting interventions for changing physical activity behaviour: a systematic review and meta-analysis. Health Psychol Rev. 2016;10(1):67-88. doi: 10.1080/17437199.2015.1104258. Epub 2015 Nov 13. PMID 26445201
- [Background] Napolitano MA, Fotheringham M, Tate D, Sciamanna C, Leslie E, Owen N, Bauman A, Marcus B. Evaluation of an internet-based physical activity intervention: a preliminary investigation. Ann Behav Med. 2003 Spring;25(2):92-9. doi: 10.1207/S15324796ABM2502_04. PMID 12704010
- [Background] Greene GW, White AA, Hoerr SL, Lohse B, Schembre SM, Riebe D, Patterson J, Kattelmann KK, Shoff S, Horacek T, Blissmer B, Phillips BW. Impact of an online healthful eating and physical activity program for college students. Am J Health Promot. 2012 Nov-Dec;27(2):e47-58. doi: 10.4278/ajhp.110606-QUAN-239. PMID 23113786
- [Background] Rovniak LS, Hovell MF, Wojcik JR, Winett RA, Martinez-Donate AP. Enhancing theoretical fidelity: an e-mail-based walking program demonstration. Am J Health Promot. 2005 Nov-Dec;20(2):85-95. doi: 10.4278/0890-1171-20.2.85. PMID 16295700
- [Background] Joseph RP, Keller C, Adams MA, Ainsworth BE. Print versus a culturally-relevant Facebook and text message delivered intervention to promote physical activity in African American women: a randomized pilot trial. BMC Womens Health. 2015 Mar 27;15:30. doi: 10.1186/s12905-015-0186-1. PMID 25886945
- [Background] Taylor WC, Paxton RJ, Shegog R, Coan SP, Dubin A, Page TF, Rempel DM. Impact of Booster Breaks and Computer Prompts on Physical Activity and Sedentary Behavior Among Desk-Based Workers: A Cluster-Randomized Controlled Trial. Prev Chronic Dis. 2016 Nov 17;13:E155. doi: 10.5888/pcd13.160231. PMID 27854422
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- See also: 2018 Physical Activity Guidelines Advisory Committee Scientific Report — https://health.gov/news-archive/blog-bayw/2018/03/2018-physical-activity-guidelines-advisory-committee-submits-scientific-report/index.html
- See also: Move Your Way Campaign — https://health.gov/our-work/physical-activity/move-your-way-campaign
- See also: Physical Activity Guidelines Figure depicting 150-minutes per week of moderate intensity aerobic physical activity plus two days of muscle strengthening activity — https://health.gov/moveyourway